CLINICAL TRIAL: NCT01793597
Title: Platelet Activation, Reactivity, and Inflammation After Coronary Bypass Surgery In Patients Treated With Ticagrelor or Clopidogrel
Brief Title: Platelet Reactivity After CABG
Status: Completed | Type: Observational
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, David J. Schneider, MD, Professor Of Medicine, Director of Cardiology, University of Vermont
Other Study IDs: ISSBRIL0095
Record Dates: First submitted 2013-02-13; First posted 2013-02-15 (Estimated); Last update posted 2015-09-22 (Estimated); Status verified 2015-09

CONDITIONS: Acute Coronary Syndrome
Keywords: ticagrelor; Coronary artery bypass surgery; platelet function; receptor binding; platelet reactivity; reversible binding
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Platelets and leukocytes will be evaluated acutely. Plasma will be stored for cytokine and chemokine analysis.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- clopidogrel: previous treatment with clopidogrel
- ticagrelor: previous treatment with ticagrelor

SUMMARY:
Patients who have a heart attack are regularly treated with either clopidogrel or ticagrelor. In a large clinical trial, treatment with ticagrelor before coronary bypass surgery (CABG) was associated with a lower risk of death than treatment with clopidogrel. The reason for this difference cannot be explained on the basis of the study. One possible explanation is that the reversible binding of ticagrelor is advantageous because when new platelets are released, they are inhibited by the drug. Because clopidogrel binds irreversibly it cannot redistribute. The investigators will recruit patients who are scheduled for surgery after an acute coronary syndrome who have been treated with either ticagrelor or clopidogrel. After the patient provides informed consent, the investigators will review their medical record,record information and on the day after surgery the investigators will take one sample of blood. That blood will be analyzed for evidence of platelet activation (platelet microparticles, and platelet-leukocyte aggregates), the reactivity of young platelets, and the concentration of inflammatory cytokines. The investigators hypothesize that the evidence of platelet activation (platelet microparticles and platelet-leukocyte aggregates) and the reactivity of young platelets will be less in patients who have been treated previously with ticagrelor.

ELIGIBILITY:
Inclusion Criteria:

* Acute coronary syndrome, CABG, within 48 hours of last dose of clopidogrel or ticagrelor, treatment with aspirin

Exclusion Criteria:

* Treatment with an antiplatelet agent other than aspirin, clopidogrel, or ticagrelor, Acute or chronic hematologic disorder including a preoperative Hgb less than 10 g/dl or platelet count less than 100,000/mm3, Moderate or severe renal insufficiency (glomerular filtration rate less than 60 ml/min), Active infection, Active malignancy, Unable/unwilling to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute coronary syndrome who based on clinical indications require urgent CABG. CABG is scheduled for clinical indications within 48 hours. Previous treatment with clopidogrel or ticagrelor.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2013-05; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
reactivity of juvenile platelets | 16-24 hours after CABG
  We will use flow cytometry to identify juvenile platelets and assess their likelihood to activate in response to a submaximal concentration of agonist.

SECONDARY OUTCOMES:
platelet-leukocyte aggregates | 16-24 hours after CABG
  We will identify the prevalence of platelet-leukocyte aggregates - a marker of platelet activation in vivo
platelet microparticles | 16-24 hours after CABG
  We will quantify the prevalence of platelet microparticles, reflecting platelet activation in vivo
cytokine/chemokine array | 16-24 hours after CABG
  We will quantify the concentration of common cytokines and chemokines.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Vermont Medical Center, Burlington, Vermont, United States